CLINICAL TRIAL: NCT03976622
Title: Analysis of Inflammation in the Vitiligo and Other Inflammatory Skin Diseases: Psoriasis, Atopic Dermatitis and Alopecia Areata
Acronym: INFLAMMAVit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/55
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Vitiligo; Psoriasis; Alopecia Areata; Atopic Dermatitis
Keywords: Skin inflammation; Cytokines
MeSH Terms: conditions — Vitiligo; Psoriasis; Alopecia Areata; Dermatitis, Atopic; Dermatitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral mononuclear cells, Serum, paraffine-embedded/ frozen skin.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- vitiligo: Patients aged 18 to 75 years with non-segmental vitiligo;
  Interventions: Biological: Blood samples; Biological: Skin biopsies
- psoriasis: Patients aged 18 to 75 years with plaque psoriasis;
  Interventions: Biological: Blood samples; Biological: Skin biopsies
- atopic dermatitis: Patients aged 18 to 75 years with atopic dermatitis;
  Interventions: Biological: Blood samples; Biological: Skin biopsies
- alopecia areata: Patients aged 18 to 75 years with alopecia areata sclerosis;
  Interventions: Biological: Blood samples; Biological: Skin biopsies

INTERVENTIONS:
Biological: Blood samples — Blood samples: serum and PBMC
  Other Names: Blood samples: serum and PBMC
Biological: Skin biopsies — These superficial skin biopsies under local anesthesia in skin areas with the exception of the face and folds.

SUMMARY:
It is a study of translational research with mechanistically objectives and including biological samples of patients with chronic inflammatory disorders

DETAILED DESCRIPTION:
This study was a single-center prospective study to collect blood and skin tissue at the time of consultation with a patient with non-segmental vitiligo, psoriasis, atopic dermatitis or alopecia areata, in order to better understand and compare blood and skin immune response in chronic inflammatory skin disorders: psoriasis, alopecia areata, atopic dermatitis and vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years;
* Patients with non-segmental vitiligo;
* Patients with plaque psoriasis;
* Patients with atopic dermatitis;
* Patients with alopecia areata sclerosis;
* written consent, free, informed and signed by the patient and the investigator (before any examination required by the study);
* Subject affiliated or beneficiary of a social security system.

Exclusion Criteria:

* Patients with segmental vitiligo
* Patients under local treatment (topical corticosteroid-Calcineurin inhibitor) for less than two weeks.
* Patients on therapy, systemic treatments: acitretin, methotrexate, cyclosporine, Apremilast, infliximab, adalimumab, etanercept, ustekinumab, secukinumab, ixekizumab, dupilumab) for less than 4 weeks.
* Pregnant or breastfeeding women
* Patient (e) under guardianship
* Patient (e) Non-affiliated (e) a social protection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 450 patients (300 patients with vitiligo, 50 psoriasis patients, 50 patients with atopic dermatitis, 50 patients with alopecia areata)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-06-03 (Estimated); Primary Completion 2023-06-03 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
Description of the phenotype and function of blood and skin T-cell in chronic inflammatory skin disorders: psoriasis, vitiligo, atopic dermatitis, alopecia areata | Day 1
  Description of the phenotypic analysis of cutaneous T-cell and blood of vitiligo patients evaluated by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Julien SENESCHAL, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Dermatologie - Hôpital Saint-André, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No